CLINICAL TRIAL: NCT06230705
Title: Community Intervention to impRove CVD Risk Factor controL in Young AmErican Indians: The CIRCLE Study
Brief Title: Community Intervention to Improve CVD Risk Factor Control in Young American Indians
Acronym: CIRCLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 118014
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cholesterol, Elevated; Diabetes Mellitus
Keywords: Elevated Cholesterol; Diabetes Mellitus; Cardiovascular Disease; American Indian; Young Adult
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus; Cardiovascular Diseases | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided management (Experimental): The intervention will be comprised of four broad components (described below). The focus groups will inform these components and therefore, we propose a community-responsive and ultimately, community-driven intervention.
  1. Component on reducing barriers to health care access
  2. Nutritional component
  3. Activity component
  4. CVD risk factor education component
  Interventions: Other: Guided management
- Self-managed (Active Comparator): Self-managed (control group): For participants randomized to the self-managed group, we will employ the standard of care that is currently used by the Strong Heart Study (SHS) and other large cohorts, which is based on a referral program for risk factor control and dissemination of educational pamphlets. Therefore, the risk factor control and education for this group will be self-managed.
  Interventions: Other: Self management

INTERVENTIONS:
Other: Guided management — Guided Management
  Arms: Guided management
Other: Self management — Self management
  Arms: Self-managed

SUMMARY:
American Indians are more likely to die from heart disease compared to other people in the United States. High levels of fat (lipids) and sugar (glucose) in the blood are related to heart disease. Young American Indians who are 18 to 39 years old have high lipid and glucose levels. This has led to heart disease later in life. This means they are likely to benefit from a program to lower these levels.

In this project, researchers will work with American Indians in rural southwestern Oklahoma. The researchers will start by asking American Indians how they would like to design a program for younger members of their community. After getting permission, the researchers will take a small amount of blood from young community members. The researchers will measure lipid and glucose levels and ask those with high levels to be in the study. Then the researchers will do several measurements. These will include blood pressure, height, weight, diet, physical activity, sleep, tobacco and alcohol use, access to health care, and social support. The researchers will compare these measurements to similar measurements taken from young American Indians 20 years ago, collected through the Strong Heart Study, which is the longest running study measuring heart disease in American Indians.

Next, the researchers want to know if the program they developed with the American Indian communities will work. To do this, they will put people in one of two groups. They will decide which group each person will be in using a process that is like flipping a coin (heads for one group, tails for the other group). One group will receive educational booklets about how to avoid getting heart disease. The other group will receive help from a community health worker. The community health worker will help participants to get to the doctor for treatment. They will also help participants change their diet and exercise routines and provide education about heart disease risk factors. After 9 and 18 months, the researchers will repeat the measurements to see if one of the groups has lower lipid or glucose levels.

This program will support the National Heart, Lung, and Blood Institute's mission to "reduce human disease" by lowering lipid and glucose levels, which are related to getting heart disease. This will be done by using the community health worker model to help people go to the doctor and improve their lifestyle related to diet and exercise. The researchers will also be able to advance heart health in American Indians in rural Oklahoma by lowering factors related to heart disease.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) incidence in American Indians is more than two-fold higher than the age-matched United States (US) population, and significantly associated with elevated lipids/lipoproteins and glucose levels. Through systematic surveillance conducted by the Strong Heart Study (SHS), the largest and longest running study of CVD in American Indians, we report that elevated lipid/lipoprotein prevalence for participants <20, 20-29, and 30-39 years old was 55.2%, 73.6%, and 78.0%, respectively. In addition, we report that American Indians under 40 years old with elevated LDL cholesterol had a three-fold greater independent risk of subclinical atherosclerosis five (5) years later and/or incident, clinical CVD 20 years later. Although statin therapy is effective for dyslipidemia, the rates of use are low among American Indians, with less than 50% of young SHS participants with primary hypercholesterolemia receiving treatment. In addition, the high diabetes prevalence (8%) in young American Indians contributes to high rates of CVD, where incidence of atherosclerosis was 41.3 per 1,000 person-years in diabetics compared to 16.3 per 1,000 person-years in non-diabetics (p<0.001). These elevated lipid/lipoprotein and glucose levels may be due to limited health care access and lifestyle factors such as nutrition, physical activity, sleep hygiene, and social determinants of health (SDOH), including social support. As a result, there is a critical need to measure these factors and include them in a culturally appropriate intervention to control lipid/lipoprotein and glucose levels and thereby reduce CVD.

The long-term goal of this research, which aligns with the NHLBI's strategic goal to "reduce human disease," is to reduce incident CVD risk in American Indians. Our overall objective is to determine the effectiveness of a culturally appropriate intervention, designed with American Indian involvement, to control lipid/lipoprotein and glucose levels. To achieve this objective, we will determine the effectiveness of a guided intervention. Before determining the intervention effectiveness, we will use a community-engaged approach and conduct focus groups asking participants to offer recommendations for a modified version of the Balance Study that we conducted with older (mean age=52 years) American Indians in Oklahoma, 2008-2012. Subsequently, we will recruit 360 American Indians, 18-39 years old, with elevated lipid/lipoprotein or glucose levels. Among this group, we will assess baseline CVD risk factors and then randomly assign them to either a self-managed control group receiving health care referrals and educational materials or to an 18-month guided intervention group, incorporating: 1) community health workers (CHW) to reduce health care access barriers and 2) a multidimensional component focusing on nutrition, physical activity, and CVD risk factor education during at least six (6) quarterly in-person meetings. Based on the Balance Study and SHS, we formulated the central hypothesis that health care access, nutrition, physical activity, and CVD risk factor education jointly contribute to lipid/lipoprotein and glucose control. Therefore, the rationale for the proposed research is to include these components in an intervention targeting lipid/lipoprotein and glucose management. Given our experience with American Indian communities recruiting and designing interventions for the SHS, we are well-positioned to conduct this research, with the following Specific Aims:

Aim 1: (A) To work with CHWs, healthcare workers, community leaders, and community members to adapt a culturally relevant CVD risk factor intervention based on the Balance Study for American Indians, 18-39 years old. (B) To assess the acceptability of the adapted intervention among American Indians, 18-39 years old from communities participating in the Strong Heart Study in southwestern Oklahoma. We will work with members of the community to adapt a lifestyle intervention for younger populations that was previously used in older populations of American Indians, titled the Balance Study. Then we will conduct focus groups among American Indians who are 18-29 or 30-39 to determine the acceptability of adapted intervention among these groups.

Aim 2: To determine if the adapted 18-month guided intervention is more effective than self-management at lowering LDL-C or glucose levels, among American Indians, with serum LDL-C ≥100 mg/dL and/or fasting plasma glucose ≥126 mg/dL who are 18-39 years old from communities participating in the Strong Heart Study in southwestern Oklahoma. Hypothesis: American Indians, 18-39 years old, randomized to the guided intervention, will have at least a 10% reduction in LDL-C and/or glucose levels after 18 months.

The proposed research will determine the effectiveness of an intervention that uses the CHW model to target health care access, nutrition, physical activity, and CVD risk factor education within the young adult American Indian population. The expected outcomes include the refinement of a culturally appropriate CVD risk factor reduction intervention and the reduction of LDL-C and glucose levels in young American Indians with elevated CVD risk. This study will decrease the disproportionately high lipid/lipoprotein and glucose levels that are significantly predictive of incident CVD in young American Indians.

ELIGIBILITY:
Inclusion Criteria:

* American Indians
* 18-39 years old
* Members of the tribal communities that participate in the Strong Heart Study in southwestern Oklahoma
* Only one person per household will be eligible

Exclusion Criteria:

* Are unwilling or unable to follow the intervention, which includes modifying current nutritional intake and participating in the proposed physical activity program
* Are taking lipid-/lipoprotein-lowering or diabetes medication
* Are already participating in a diabetes or CVD risk factor reduction program
* Are pregnant or plan to become pregnant in the next 18 months
* Are not English speaking
* Are institutionalized
* Have underlying disease with a life-expectancy of less than 2 years (e.g., cancer or end stage renal disease).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Lipid Levels | 9 and 18 months
  LDL cholesterol
Glucose Levels | 9 and 18 months
  Fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Reese, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Heath Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be collected, analyzed, and reported under agreements made with the sovereign tribal nations that have partnered in this research, which preclude commonly accepted modes of data sharing. Requests will be reviewed by tribal research partners before data may be released. This policy is consistent with the "NIH Policy for Data Management and Sharing: Responsible Management and Sharing of American Indian/Alaska Native Participant Data."
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the end of the study period. Data will be available after tribal approval.
Access Criteria: Tribal approval
URL: https://grants.nih.gov/grants/guide/notice-files/NOT-OD-22-214.html

REFERENCES:
- [Background] Lee ET, Welty TK, Fabsitz R, Cowan LD, Le NA, Oopik AJ, Cucchiara AJ, Savage PJ, Howard BV. The Strong Heart Study. A study of cardiovascular disease in American Indians: design and methods. Am J Epidemiol. 1990 Dec;132(6):1141-55. doi: 10.1093/oxfordjournals.aje.a115757. PMID 2260546
- [Background] Howard BV, Lee ET, Cowan LD, Devereux RB, Galloway JM, Go OT, Howard WJ, Rhoades ER, Robbins DC, Sievers ML, Welty TK. Rising tide of cardiovascular disease in American Indians. The Strong Heart Study. Circulation. 1999 May 11;99(18):2389-95. doi: 10.1161/01.cir.99.18.2389. PMID 10318659
- [Background] Cross SH, Califf RM, Warraich HJ. Rural-Urban Disparity in Mortality in the US From 1999 to 2019. JAMA. 2021 Jun 8;325(22):2312-2314. doi: 10.1001/jama.2021.5334. PMID 34100876
- [Background] Lee ET, Cowan LD, Welty TK, Sievers M, Howard WJ, Oopik A, Wang W, Yeh J, Devereux RB, Rhoades ER, Fabsitz RR, Go O, Howard BV. All-cause mortality and cardiovascular disease mortality in three American Indian populations, aged 45-74 years, 1984-1988. The Strong Heart Study. Am J Epidemiol. 1998 Jun 1;147(11):995-1008. doi: 10.1093/oxfordjournals.aje.a009406. PMID 9620042
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Reese J, Roman MJ, Deen J, Ali T, Cole S, Devereux RB, Fretts AM, Howard BV, Howard WJ, Lee ET, et al. Abstract P040: Dyslipidemia And The Incidence Of Subclinical And Clinical Cardiovascular Disease In Adolescents And Young Adults: The Strong Heart Family Study (SHFS). Circulation. 2022;145:AP040-AP040. doi:doi:10.1161/circ.145.suppl_1.P040
- [Background] De Marco M, de Simone G, Roman MJ, Chinali M, Lee ET, Calhoun D, Howard BV, Devereux RB. Cardiac geometry and function in diabetic or prediabetic adolescents and young adults: the Strong Heart Study. Diabetes Care. 2011 Oct;34(10):2300-5. doi: 10.2337/dc11-0191. Epub 2011 Aug 26. PMID 21873564
- [Background] Lee JS, Chang PY, Zhang Y, Kizer JR, Best LG, Howard BV. Triglyceride and HDL-C Dyslipidemia and Risks of Coronary Heart Disease and Ischemic Stroke by Glycemic Dysregulation Status: The Strong Heart Study. Diabetes Care. 2017 Apr;40(4):529-537. doi: 10.2337/dc16-1958. Epub 2017 Jan 25. PMID 28122840
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):e285-e350. doi: 10.1016/j.jacc.2018.11.003. Epub 2018 Nov 10. No abstract available. PMID 30423393
- [Background] Zhang Y, Galloway JM, Welty TK, Wiebers DO, Whisnant JP, Devereux RB, Kizer JR, Howard BV, Cowan LD, Yeh J, Howard WJ, Wang W, Best L, Lee ET. Incidence and risk factors for stroke in American Indians: the Strong Heart Study. Circulation. 2008 Oct 7;118(15):1577-84. doi: 10.1161/CIRCULATIONAHA.108.772285. Epub 2008 Sep 22. PMID 18809797
- [Background] Howard BV, Roman MJ, Devereux RB, Fleg JL, Galloway JM, Henderson JA, Howard WJ, Lee ET, Mete M, Poolaw B, Ratner RE, Russell M, Silverman A, Stylianou M, Umans JG, Wang W, Weir MR, Weissman NJ, Wilson C, Yeh F, Zhu J. Effect of lower targets for blood pressure and LDL cholesterol on atherosclerosis in diabetes: the SANDS randomized trial. JAMA. 2008 Apr 9;299(14):1678-89. doi: 10.1001/jama.299.14.1678. PMID 18398080
- [Background] Howard WJ, Russell M, Fleg JL, Mete M, Ali T, Devereux RB, Galloway JM, Otvos JD, Ratner RE, Roman MJ, Silverman A, Umans JG, Weissman NJ, Wilson C, Howard BV. PREVENTION OF ATHEROSCLEROSIS WITH LDL-C LOWERING - LIPOPROTEIN CHANGES AND INTERACTIONS: THE SANDS STUDY. J Clin Lipidol. 2009 Oct 1;3(5):322-331. doi: 10.1016/j.jacl.2009.09.001. PMID 20161568
- [Background] de Simone G, Devereux RB, Chinali M, Best LG, Lee ET, Galloway JM, Resnick HE; Strong Heart Study Investigators. Prognostic impact of metabolic syndrome by different definitions in a population with high prevalence of obesity and diabetes: the Strong Heart Study. Diabetes Care. 2007 Jul;30(7):1851-6. doi: 10.2337/dc06-2152. Epub 2007 Apr 17. PMID 17440172
- [Background] Reese JA, Roman MJ, Deen JF, Ali T, Cole SA, Devereux RB, Fretts AM, Howard BV, Lee ET, Malloy K, Singh P, Umans JG, Zhang Y. Subclinical atherosclerosis in adolescents and young adults and the risk of cardiovascular disease: The Strong Heart Family Study (SHFS). Nutr Metab Cardiovasc Dis. 2022 Aug;32(8):1863-1871. doi: 10.1016/j.numecd.2022.04.024. Epub 2022 May 10. PMID 35680485
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027
- [Background] Balcazar H, Wise S, Rosenthal EL, Ochoa C, Rodriguez J, Hastings D, Flores L, Hernandez L, Duarte-Gardea M. An ecological model using promotores de salud to prevent cardiovascular disease on the US-Mexico border: the HEART project. Prev Chronic Dis. 2012;9:E35. doi: 10.5888/pcd9.110100. Epub 2012 Jan 12. PMID 22239750
- [Background] Jernigan V, Lee ET, Yeh J, Fabsitz RR, Howard BV and Zhang Y. Abstract P373: Health Care Access and Usage Patterns Among Native Americans: The Strong Heart Study. Circulation. 2023;147:AP373-AP373. doi:doi:10.1161/circ.147.suppl_1.P373.
- [Background] Kauffman SAE, Averill MM, Delaney JAC, Lemaitre RN, Howard BV, Fretts AM. Associations of diet quality and blood serum lipoprotein levels in a population at high risk for diabetes: the Strong Heart Family Study. Eur J Clin Nutr. 2020 Jul;74(7):1084-1090. doi: 10.1038/s41430-019-0539-1. Epub 2019 Dec 5. PMID 31804627
- [Background] Suchy-Dicey AM, Vo TT, Oziel K, King R, Barbosa-Leiker C, Rhoads K, Verney S, Buchwald DS, French BF. Psychometric Properties of Controlled Oral Word Association (COWA) Test and Associations With Education and Bilingualism in American Indian Adults: The Strong Heart Study. Assessment. 2024 Apr;31(3):745-757. doi: 10.1177/10731911231180127. Epub 2023 Jun 20. PMID 37338127
- [Background] Suchy-Dicey A, Eyituoyo H, O'Leary M, Cole SA, Traore A, Verney S, Howard B, Manson S, Buchwald D, Whitney P. Psychological and social support associations with mortality and cardiovascular disease in middle-aged American Indians: the Strong Heart Study. Soc Psychiatry Psychiatr Epidemiol. 2022 Jul;57(7):1421-1433. doi: 10.1007/s00127-022-02237-7. Epub 2022 Feb 14. PMID 35157091
- [Background] Oetzel J, Duran B, Jiang Y, Lucero J. Social support and social undermining as correlates for alcohol, drug, and mental disorders in American Indian women presenting for primary care at an Indian Health Service hospital. J Health Commun. 2007 Mar;12(2):187-206. doi: 10.1080/10810730601152771. PMID 17365359
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Beals J, Manson SM, Mitchell CM, Spicer P; AI-SUPERPFP Team. Cultural specificity and comparison in psychiatric epidemiology: walking the tightrope in American Indian research. Cult Med Psychiatry. 2003 Sep;27(3):259-89. doi: 10.1023/a:1025347130953. PMID 14510095
- [Background] Stokols D. Translating social ecological theory into guidelines for community health promotion. Am J Health Promot. 1996 Mar-Apr;10(4):282-98. doi: 10.4278/0890-1171-10.4.282. PMID 10159709
- [Background] Lee ET, Jobe JB, Yeh J, Ali T, Rhoades ER, Knehans AW, Willis DJ, Johnson MR, Zhang Y, Poolaw B, Rogers B. A cardiovascular risk reduction program for American Indians with metabolic syndrome: the Balance Study. J Prim Prev. 2012 Aug;33(4):187-96. doi: 10.1007/s10935-012-0273-0. PMID 22941041
- [Background] Banna J, Bersamin A. Community involvement in design, implementation and evaluation of nutrition interventions to reduce chronic diseases in indigenous populations in the U.S.: a systematic review. Int J Equity Health. 2018 Aug 13;17(1):116. doi: 10.1186/s12939-018-0829-6. PMID 30103753
- [Background] Lee ET, Begum M, Wang W, Blackett PR, Blevins KS, Stoddart M, Tolbert B, Alaupovic P. Type 2 diabetes and impaired fasting glucose in American Indians aged 5-40 years: the Cherokee diabetes study. Ann Epidemiol. 2004 Oct;14(9):696-704. doi: 10.1016/j.annepidem.2003.10.013. PMID 15380801
- [Background] Noe TD, Manson SM, Croy C, McGough H, Henderson JA, Buchwald DS. The influence of community-based participatory research principles on the likelihood of participation in health research in American Indian communities. Ethn Dis. 2007 Winter;17(1 Suppl 1):S6-14. PMID 17598311
- [Background] Wallerstein NB, Duran B. Using community-based participatory research to address health disparities. Health Promot Pract. 2006 Jul;7(3):312-23. doi: 10.1177/1524839906289376. Epub 2006 Jun 7. PMID 16760238
- [Background] Chinali M, de Simone G, Roman MJ, Best LG, Lee ET, Russell M, Howard BV, Devereux RB. Cardiac markers of pre-clinical disease in adolescents with the metabolic syndrome: the strong heart study. J Am Coll Cardiol. 2008 Sep 9;52(11):932-8. doi: 10.1016/j.jacc.2008.04.013. PMID 18772065
- [Background] Bucholz EM, Gooding HC, de Ferranti SD. Awareness of Cardiovascular Risk Factors in U.S. Young Adults Aged 18-39 Years. Am J Prev Med. 2018 Apr;54(4):e67-e77. doi: 10.1016/j.amepre.2018.01.022. Epub 2018 Feb 9. PMID 29433955
- [Background] Sturlaugsdottir R, Aspelund T, Bjornsdottir G, Sigurdsson S, Thorsson B, Eiriksdottir G, Gudnason V. Prevalence and determinants of carotid plaque in the cross-sectional REFINE-Reykjavik study. BMJ Open. 2016 Nov 24;6(11):e012457. doi: 10.1136/bmjopen-2016-012457. PMID 27884845
- [Background] Russell M, Fleg JL, Galloway WJ, Henderson JA, Howard J, Lee ET, Poolaw B, Ratner RE, Roman MJ, Silverman A, Stylianou M, Weir MR, Wilson C, Yeh F, Zhu J, Howard BV. Examination of lower targets for low-density lipoprotein cholesterol and blood pressure in diabetes--the Stop Atherosclerosis in Native Diabetics Study (SANDS). Am Heart J. 2006 Nov;152(5):867-75. doi: 10.1016/j.ahj.2006.05.021. PMID 17070147
- [Background] Wagner J, Lacey K, Chyun D, Abbott G. Development of a questionnaire to measure heart disease risk knowledge in people with diabetes: the Heart Disease Fact Questionnaire. Patient Educ Couns. 2005 Jul;58(1):82-7. doi: 10.1016/j.pec.2004.07.004. PMID 15950840
- [Background] Eisele M, Reese J, Jones A and Zhang Y. Abstract P646: American Indian Community Stakeholders Evaluate the Cardiovascular Health Curriculum Honoring the Gift of Heart Health: The Strong Heart Study. Circulation. 2023;147:AP646-AP646. doi:doi:10.1161/circ.147.suppl_1.P646.
- [Background] North KE, Howard BV, Welty TK, Best LG, Lee ET, Yeh JL, Fabsitz RR, Roman MJ, MacCluer JW. Genetic and environmental contributions to cardiovascular disease risk in American Indians: the strong heart family study. Am J Epidemiol. 2003 Feb 15;157(4):303-14. doi: 10.1093/aje/kwf208. PMID 12578801
- [Background] Stoddart ML, Jarvis B, Blake B, Fabsitz RR, Howard BV, Lee ET, Welty TK. Recruitment of American Indians in epidemiologic research: the Strong Heart Study. Am Indian Alsk Native Ment Health Res. 2000;9(3):20-37. doi: 10.5820/aian.0903.2000.20. PMID 11279560
- [Background] Triplett C, Fletcher BJ, Taitingfong RI, Zhang Y, Ali T, Ohno-Machado L, Bloss CS. Codesigning a community-based participatory research project to assess tribal perspectives on privacy and health data sharing: A report from the Strong Heart Study. J Am Med Inform Assoc. 2022 May 11;29(6):1120-1127. doi: 10.1093/jamia/ocac038. PMID 35349678
- [Background] Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: assessing partnership approaches to improve public health. Annu Rev Public Health. 1998;19:173-202. doi: 10.1146/annurev.publhealth.19.1.173. PMID 9611617
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Brega AG, Pratte KA, Jiang L, Mitchell CM, Stotz SA, Loudhawk-Hedgepeth C, Morse BD, Noe T, Moore KR, Beals J. Impact of targeted health promotion on cardiovascular knowledge among American Indians and Alaska Natives. Health Educ Res. 2013 Jun;28(3):437-49. doi: 10.1093/her/cyt054. PMID 23660462
- [Background] Rogers EJ, Misner L, Ockene IS, Nicolosi RJ. Evaluation of seven Cholestech L.D.X analyzers for total cholesterol determinations. Clin Chem. 1993 May;39(5):860-4. PMID 8485877
- [Background] Roman MJ, Kizer JR, Best LG, Lee ET, Howard BV, Shara NM, Devereux RB. Vascular biomarkers in the prediction of clinical cardiovascular disease: the Strong Heart Study. Hypertension. 2012 Jan;59(1):29-35. doi: 10.1161/HYPERTENSIONAHA.111.181925. Epub 2011 Nov 7. PMID 22068872
- [Background] Halpern A, Mancini MC, Magalhaes ME, Fisberg M, Radominski R, Bertolami MC, Bertolami A, de Melo ME, Zanella MT, Queiroz MS, Nery M. Metabolic syndrome, dyslipidemia, hypertension and type 2 diabetes in youth: from diagnosis to treatment. Diabetol Metab Syndr. 2010 Aug 18;2:55. doi: 10.1186/1758-5996-2-55. PMID 20718958
- [Background] Drukteinis JS, Roman MJ, Fabsitz RR, Lee ET, Best LG, Russell M, Devereux RB. Cardiac and systemic hemodynamic characteristics of hypertension and prehypertension in adolescents and young adults: the Strong Heart Study. Circulation. 2007 Jan 16;115(2):221-7. doi: 10.1161/CIRCULATIONAHA.106.668921. Epub 2007 Jan 8. PMID 17210838
- [Background] Zhang M, An Q, Yeh F, Zhang Y, Howard BV, Lee ET, Zhao J. Smoking-attributable mortality in American Indians: findings from the Strong Heart Study. Eur J Epidemiol. 2015 Jul;30(7):553-61. doi: 10.1007/s10654-015-0031-8. Epub 2015 May 13. PMID 25968176
- [Background] Lowe LP, Long CR, Wallace RB, Welty TK. Epidemiology of alcohol use in a group of older American Indians. Ann Epidemiol. 1997 May;7(4):241-8. doi: 10.1016/s1047-2797(97)00003-3. PMID 9177105
- [Background] Block G, Thompson FE, Hartman AM, Larkin FA, Guire KE. Comparison of two dietary questionnaires validated against multiple dietary records collected during a 1-year period. J Am Diet Assoc. 1992 Jun;92(6):686-93. PMID 1607564
- [Background] Caan BJ, Slattery ML, Potter J, Quesenberry CP Jr, Coates AO, Schaffer DM. Comparison of the Block and the Willett self-administered semiquantitative food frequency questionnaires with an interviewer-administered dietary history. Am J Epidemiol. 1998 Dec 15;148(12):1137-47. doi: 10.1093/oxfordjournals.aje.a009598. PMID 9867257
- [Background] Santos RMGD, De Martino JM, Haiter Neto F, Passeri LA. Influence of different setups of the Frankfort horizontal plane on 3-dimensional cephalometric measurements. Am J Orthod Dentofacial Orthop. 2017 Aug;152(2):242-249. doi: 10.1016/j.ajodo.2016.12.023. PMID 28760286
- [Background] Chinali M, de Simone G, Roman MJ, Lee ET, Best LG, Howard BV, Devereux RB. Impact of obesity on cardiac geometry and function in a population of adolescents: the Strong Heart Study. J Am Coll Cardiol. 2006 Jun 6;47(11):2267-73. doi: 10.1016/j.jacc.2006.03.004. PMID 16750694
- [Background] Gal R, May AM, van Overmeeren EJ, Simons M, Monninkhof EM. The Effect of Physical Activity Interventions Comprising Wearables and Smartphone Applications on Physical Activity: a Systematic Review and Meta-analysis. Sports Med Open. 2018 Sep 3;4(1):42. doi: 10.1186/s40798-018-0157-9. PMID 30178072
- [Background] Rhodes RE, Guerrero MD, Vanderloo LM, Barbeau K, Birken CS, Chaput JP, Faulkner G, Janssen I, Madigan S, Masse LC, McHugh TL, Perdew M, Stone K, Shelley J, Spinks N, Tamminen KA, Tomasone JR, Ward H, Welsh F, Tremblay MS. Development of a consensus statement on the role of the family in the physical activity, sedentary, and sleep behaviours of children and youth. Int J Behav Nutr Phys Act. 2020 Jun 16;17(1):74. doi: 10.1186/s12966-020-00973-0. PMID 32539730
- [Background] Andersen LB, Harro M, Sardinha LB, Froberg K, Ekelund U, Brage S, Anderssen SA. Physical activity and clustered cardiovascular risk in children: a cross-sectional study (The European Youth Heart Study). Lancet. 2006 Jul 22;368(9532):299-304. doi: 10.1016/S0140-6736(06)69075-2. PMID 16860699
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Kerr J, Rosenberg D, Millstein RA, Bolling K, Crist K, Takemoto M, Godbole S, Moran K, Natarajan L, Castro-Sweet C, Buchner D. Cluster randomized controlled trial of a multilevel physical activity intervention for older adults. Int J Behav Nutr Phys Act. 2018 Apr 2;15(1):32. doi: 10.1186/s12966-018-0658-4. PMID 29609594
- [Background] Wei LJ, Lachin JM. Properties of the urn randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):345-64. doi: 10.1016/0197-2456(88)90048-7. PMID 3203525
- [Background] Block G, Mandel R, Gold E. On food frequency questionnaires: the contribution of open-ended questions and questions on ethnic foods. Epidemiology. 2004 Mar;15(2):216-21. doi: 10.1097/01.ede.0000112144.77106.bf. PMID 15127915
- See also: Strong Heart Study Website — https://strongheartstudy.org/